CLINICAL TRIAL: NCT03795233
Title: Fecal Microbiota Transplant (FMT) After Treatment for a First Episode of Clostridium Difficile Infection (CDI)
Brief Title: Fecal Microbiota Transplant for Primary CDI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated after a covid-related suspension and the unavailability of drug.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37574
Record Dates: First submitted 2018-11-21; First posted 2019-01-07 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Clostridium Difficile Infection
Keywords: Fecal Microbiota Transplant (FMT); Vancomycin; Dysbiosis; fecal microbiome; C difficile infection
MeSH Terms: conditions — Clostridium Infections; Dysbiosis | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (Experimental): Fecal microbiota transplant G3 capsules will be administered after standard of care with oral vancomycin therapy in participants with primary Clostridium difficile infection.
  Interventions: Biological: Fecal microbiota transplant G3 capsules
- Oral vancomycin alone (Control) (Active Comparator): Oral vancomycin therapy will be administered as per standard of care in participants with primary clostridium difficile infection.
  Interventions: Other: Oral Vancomycin alone

INTERVENTIONS:
Biological: Fecal microbiota transplant G3 capsules — After standard of care therapy with oral vancomycin, frozen oral FMT capsules will be provided in a formulation designed to deliver the product to the large intestine. 30 FMT capsules will be administered over a 2 hour period under direct observation
  Other Names: FMT
  Arms: Fecal microbiota transplantation
Other: Oral Vancomycin alone — Standard of care will be provided with oral vancomycin therapy.
  Other Names: Oral Vancocin alone
  Arms: Oral vancomycin alone (Control)

SUMMARY:
Clostridium difficile infection (CDI) is one of the most urgent health threats in the U.S. associated with antibiotic use. After an initial episode, disease recurrence is high and relapses can occur in 20-30% of people treated with oral vancomycin. An antibiotic course can affect the gut microbiome for years, and patients with CDI have additional dysbiosis of their gut flora. Oral vancomycin perturbs the gut microbiome further. Restoration of the microbiome with Fecal Microbiota Transplant (FMT) has been proven a highly efficacious and cost-effective treatment for recurrent CDI. FMT has had very limited study for a primary episode of CDI to date because an endoscopic procedure was the recommended route of delivery. However, FMT is now available via frozen oral capsules and has been shown to be non-inferior to FMT via colonoscopy in randomized controlled trials.

The investigators hypothesize that outcomes after a first episode of CDI can be improved if the microbiome is restored with oral FMT. It is further hypothesized that this will compensate for any additional microbiome perturbation caused by administration of oral vancomycin and decrease the likelihood of recurrence. Because the hypothesis is based on restoration of the microbiome, the investigators propose this proof-of-concept pilot study to examine whether FMT administered after oral vancomycin therapy for primary CDI restores microbiome diversity compared to patients who do not receive FMT. Because of the potential health benefits, this approach deserves further study. The results from this pilot study on the microbiome diversity as well as the surveys to be conducted about GI symptomatology (e.g., diarrhea, abdominal pain, bloating), CDI recurrence and healthcare utilization, would provide preliminary data to support a randomized controlled, multicenter clinical trial.

DETAILED DESCRIPTION:
Population: Patients >= 18 years hospitalized at Boston Medical Center (BMC) with a first documented episode of CDI.

Intervention: 30 FMT capsules administered orally under direct observation within 7 days of completion of 10-14 day treatment of oral vancomycin for CDI.

Objectives:

1. To characterize the microbial diversity in stool samples from subjects with a primary episode of CDI before and after oral vancomycin and determine the impact of FMT after completion of oral vancomycin course.
2. To characterize the feasibility and tolerability of FMT after completion of a course of oral vancomycin therapy for primary CDI, and to describe 30-day hospital readmission and gastrointestinal symptomatology and/or CDI recurrence during 60-day follow-up.

Design/Methodology:

15 subjects will be enrolled who are hospitalized at BMC for a primary episode of CDI. A discard aliquot from baseline stool samples obtained clinically for diagnosis will be frozen. Subjects will receive the standard of care treatment (oral vancomycin for 10-14 days) and within 7 days following completion will receive oral FMT during a 2 hour visit in the Infectious Disease (ID) Clinical Trials Unit. An additional 5 subjects will be enrolled as controls. Stool samples will be collected at time of CDI diagnosis and again 3 weeks after FMT for intervention group and 4 weeks after completion of oral vancomycin treatment for control subjects. The post-treatment samples will be obtained by the patient using special stool sample collection kits known as RNAlater kits (ribonucleic acid stabilization). These contain a liquid nontoxic tissue storage reagent known as RNAlater and helps preserve the stool sample. The subjects will mail this stool sample to the BMC Clinical Trials Unit (CTU) where it will aliquoted, centrifuged and frozen.

Samples will be processed at a collaborating lab at Tufts to characterize the fecal microbiome pre- and post oral FMT.

Study personnel will contact participants via telephone 60 days after FMT dosing to administer a follow-up survey (including questions on residual symptoms. CDI recurrence, re-hospitalization, adverse events and FMT acceptability).

Total Study Duration: Anticipated time: 12 months

Subject Participation Duration: The researchers anticipate a period of 1-2 hours while an inpatient for the screening and consent process, 2 hours for the CTU visit for FMT and 20-30 minutes responding to a follow up telephone survey. Total time in the study from enrollment to completion of follow-up will be approximately 3 months and will include 10-14 days of CDI treatment with oral vancomycin (per standard of care treatment), the FMT administration and a 60 day follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary clostridium difficile infection (CDI) defined by the presence of diarrhea and a positive C. difficile Polymerase chain reaction (PCR) test
* Admitted to Boston Medical Center
* English speaking

Exclusion Criteria:

* Primary CDI treatment failure
* History of CDI
* Diagnosis of inflammatory bowel disease, immunocompromised state, or active malignancy
* Dysphagia: oropharyngeal, esophageal, functional, neuromuscular (e.g. stroke, multiple sclerosis, ALS), or patient shows evidence of dysphagia when the 'safety test' capsule is administered
* History of aspiration
* History of gastroparesis
* History of intestinal obstruction
* Severe food allergy (e.g. anaphylaxis or anaphylactoid reaction) Adverse event attributable to a previous FMT
* Patients with allergies to sodium chloride, glycerol, theobroma oil, hide bovine gelatin, sodium lauryl sulfate, Food, Drugs & Cosmetics certified colorants (FD&C), or titanium dioxide, all ingredients Generally Recognized As Safe (GRAS)
* History of ongoing antibiotic use (e.g. nitrofurantoin for urinary tract infection (UTI) prophylaxis) Currently pregnant or breastfeeding -Any condition for which the treating physician thinks the treatment may pose a health risk (e.g. severely immunocompromised)-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Barlam, MD MSC, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiota Transplantation: Fecal microbiota transplant (FMT) G3 capsules will be administered after standard of care with oral vancomycin therapy in participants with primary Clostridium difficile infection.
  Fecal microbiota transplant G3 capsules: After standard of care therapy with oral vancomycin, frozen oral FMT capsules will be provided in a formulation designed to deliver the product to the large intestine. 30 FMT capsules will be administered over a 2 hour period under direct observation
Period: Overall Study
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control) | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.9) | 58 | 51.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African Am | 2 | 0 | 2
  White | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Stool Microbiome With and Without FMT Administration
Description: The stool microbiome in participants who receive additional FMT at end of Clostridium difficile infection (CDI) treatment with oral vancomycin will be compared to the stool microbiome in participants with standard treatment or oral vancomycin alone
Time Frame: 11 months
Population: This outcome measure was not obtained on any of the participants as no participant was in the study at 11 months.
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Feasibility of Administering FMT After Completion of a Course of Oral Vancomycin Therapy
Description: The number and proportion of FMT pills participants ingest after completion of a course of oral vancomycin therapy will be documented.
Time Frame: 12 months
Population: This outcome measure was not obtained on any of the participants as no participant was in the study at 12 months.
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of FMT After a Course of Oral Vancomycin Therapy
Description: Study participants will be monitored for any adverse events to FMT such as nausea or vomiting, abdominal pain or diarrhea.
Time Frame: During test dose, during 90 minutes of FMT administration, 30 minutes after FMT administration, 48-72 hours after FMT administration
Population: Only one participant in the FMT arm ingested the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 1 | 0
Participants | 0 |

4. Secondary Outcome: Incidence of Gastrointestinal Symptomatology Based on a Survey After CDI
Description: A detailed survey with 15 questions will be administered on GI symptoms Physicians will go over any significant adverse events to determine if they are related, possibly related or unrelated to oral FMT administration
Time Frame: 60 days
Population: This outcome measure was not obtained on any of the participants.
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: CDI Recurrence
Description: Patients will be monitored for recurrent C difficile infection defined as non-resolution or recurrence of GI symptoms (abdominal pain, diarrhea etc) and/or a positive stool C difficile test The proportion of participants with CDI recurrence will be documented.
Time Frame: 60 days
Population: This outcome measure was not obtained on any of the participants.
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Hospital Readmissions After Treatment
Description: The number of hospital readmissions within 30 days after CDI treatment per patient history and chart review will be obtained
Time Frame: 30 days
Population: This outcome measure was not obtained on any of the participants.
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fecal Microbiota Transplantation | Oral Vancomycin Alone (Control)
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated after a covid-related suspension and the unavailability of drug. Data were not collected for 5 of the 6 outcomes measures and no data were collected for the primary outcome measure as no participant was in the study at the timeframe of 11 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03795233/Prot_SAP_000.pdf